CLINICAL TRIAL: NCT04213040
Title: Is Procalcitonin a Valuable Marker for the Identification of Postoperative Complications After Open-heart Surgery With Cardiopulmonary Bypass?
Brief Title: Procalcitonin and Postoperative Outcome After Open-heart Surgery
Status: Completed | Type: Observational
Sponsor: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Baysal, Associate Professor, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Other Study IDs: 2013.3/11
Record Dates: First submitted 2019-12-01; First posted 2019-12-30 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Open Heart Surgery; Cardiopulmonary Bypass; Procalcitonin; C-reactive Protein; Lactate; Outcome; Postoperative Complications
Keywords: Open heart surgery; Cardiopulmonary bypass; Procalcitonin; C-reactive protein; Lactate; Outcome; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Open-Heart Surgery for a six months duration: In a single group of patients including 146 patients undergoing openheart surgery during a period of six months, the collected parameters include; serum levels of procalcitonin, C-reactive protein, and lactate as well as postoperative complications and after this, depending on the development of postoperative complications or not in the intensive care unit patients were divided into two groups. The Group Without Complications, n=112, includes patients without a postoperative complication after open-heart surgery with cardiopulmonary bypass. The Group With Complications, n=34, includes patients with a postoperative complication after open-heart surgery with cardiopulmonary bypass.
  Interventions: Diagnostic Test: Serum levels of Procalcitonin, C-reactive protein, lactate

INTERVENTIONS:
Diagnostic Test: Serum levels of Procalcitonin, C-reactive protein, lactate — Serum PCT, CRP, and lactate values were collected postoperatively every day starting on postoperative 12 hours, postoperative days 1 through 5.
  After the operation, all postoperative complications were recorded during the first seven days period.
  The relations between diagnostic tests and postoperative complications are sought by the use of the statistical analysis methods.
  Other Names: Postoperative complications; Type of open-heart surgical operation (coronary artery bypass graft operation, mitral valve, aortic valve or multiple valvular surgeries)

SUMMARY:
The aim of this study was to investigate the impact of serum values of procalcitonin (PCT), C-reactive protein (CRP) and lactate to predict postoperative complications in the early postoperative period after open-heart surgery with cardiopulmonary bypass (CPB).

DETAILED DESCRIPTION:
The cardiopulmonary bypass (CPB) causes an inflammatory response secondary to the activation of cytokine systems in the whole body. The causes of this inflammation have been discussed extensively in the literature. As a concise summary the causes can be listed as; 1- the surgical stress, 2- the recognition of bypass circuit as an artificial surface by the blood components, 3- ischemia-reperfusion injury, 4- endotoxemia. After open-heart surgery with CPB, the development of several postoperative complications including myocardial dysfunction, respiratory failure, renal and neurologic dysfunction, bleeding disorders, altered liver function, and, multiple organ failure has been demonstrated to be related to the inflammatory response. Procalcitonin (PCT), is a 116-amino-acid protein that is produced in the liver and peripheral mononuclear cells and the normal serum PCT value is below 0.1 ng/mL in patients without signs of systemic inflammation. Serum PCT levels increase postoperatively after open-heart surgery and a peak level of 0.5 to 7.0 ng/mL is reported at 24 hours after the operation and serum PCT values decrease to normal values within seven days.

Serum C-reactive protein (CRP) values are often abnormally elevated after open-heart surgery as a result of an inflammatory response and it has not been found to be a useful prognostic marker due to its prolonged elevation after cardiac surgeries. In the literature, there are studies showing that serum PCT levels are consistently higher in patients with postoperative complications, however, a cutoff point for serum PCT to determine the risk of possible poor outcome has not been well studied. A recent study demonstrated that after CPB, serum PCT increased in patients with poor outcome especially in those who developed renal and hepatic dysfunction in addition to respiratory and circulatory insufficiency. This study demonstrated a cut off value of 2 ng/mL to predict postoperative complications. In another study, a PCT level of 2.8 ng/mL was found to be a cut off value to predict 28-day mortality in patients after coronary artery bypass grafting (CABG) however, it has been pointed out that there is a need for further studies.

The aim of our study was to investigate a relation between serum values of CRP, PCT, and lactate and development of postoperative complications (circulatory failure, pneumonia, respiratory insufficiency, sepsis, reoperation, hemorrhage, tamponade, need of inotropic support, myocardial infarction, acute kidney injury), in patients undergoing open-heart surgery with CPB. A sample size of 72 patients would have a power (1-ß) of 80% to detect a difference in serum PCT level of 10% (1 standard deviation) difference between patients with postoperative complications (n=36) and without postoperative complications (n=36) using 2-sided significance and an α=0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 and younger than 80 years old,
2. Elective open heart surgery with cardiopulmonary bypass (CPB),
3. American Society of Anesthesiology (ASA) physical status of 2 or 3.

Exclusion Criteria:

1. Perioperative signs of infection (preoperatively, during operation or postoperatively during the study period) including a report of fever greater than 38 degrees centigrade, increase in white blood cell count, increase in C-reactive protein value,
2. The detection of pneumonia including infiltration in chest x-ray,
3. The diagnosis of multiple organ failure,
4. The use of corticosteroids or non-steroidal anti-inflammatory drugs within the last seven days before surgery.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is performed on a patient population undergoing open-heart surgery with cardiopulmonary bypass.
Sampling Method: Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2013-07-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
The comparison of serum procalcitonin values postoperatively | Postoperatively every day starting on postoperative 12 hours, postoperative days 1 through 5.
  Serum Procalcitonin values were collected postoperatively for five days and a change from the postoperative 12 hours value was evaluated using appropriate statistical analysis. Later, a repeated measures statistical analysis was also performed.
The comparison of serum-reactive protein values postoperatively | Postoperatively every day starting on postoperative 12 hours, postoperative days 1 through 5.
  Serum C-reactive protein values were collected postoperatively for five days and a change from the postoperative 12 hours value was evaluated using appropriate statistical analysis. Later, a repeated measures statistical analysis was also performed.
The comparison of serum lactate values postoperatively | Postoperatively every day starting on postoperative 12 hours, postoperative days 1 through 5.
  Serum Lactate values were collected postoperatively for five days and a change from the postoperative 12 hours value was evaluated using appropriate statistical analysis. Later, a repeated measures statistical analysis was also performed.

SECONDARY OUTCOMES:
Complications | Postoperatively for a duration of seven days after operation.
  Postoperative complications were collected and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Baysal, MD, Principal Investigator — Pendik Bolge Hospital

IPD SHARING:
Plan to Share IPD: Yes
We can share the study protocol, clinical study report, the excel and spss data of our clinical work.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data is available upon registration and it will be available in the web site if needed.
Access Criteria: Accessible to all researchers.

REFERENCES:
- [Background] Warren OJ, Smith AJ, Alexiou C, Rogers PL, Jawad N, Vincent C, Darzi AW, Athanasiou T. The inflammatory response to cardiopulmonary bypass: part 1--mechanisms of pathogenesis. J Cardiothorac Vasc Anesth. 2009 Apr;23(2):223-31. doi: 10.1053/j.jvca.2008.08.007. Epub 2008 Oct 19. No abstract available. PMID 18930659
- [Background] Vohra HA, Whistance R, Modi A, Ohri SK. The inflammatory response to miniaturised extracorporeal circulation: a review of the literature. Mediators Inflamm. 2009;2009:707042. doi: 10.1155/2009/707042. Epub 2010 Jan 13. PMID 20101278
- [Result] Sponholz C, Sakr Y, Reinhart K, Brunkhorst F. Diagnostic value and prognostic implications of serum procalcitonin after cardiac surgery: a systematic review of the literature. Crit Care. 2006;10(5):R145. doi: 10.1186/cc5067. PMID 17038199
- [Result] Aouifi A, Piriou V, Blanc P, Bouvier H, Bastien O, Chiari P, Rousson R, Evans R, Lehot JJ. Effect of cardiopulmonary bypass on serum procalcitonin and C-reactive protein concentrations. Br J Anaesth. 1999 Oct;83(4):602-7. doi: 10.1093/bja/83.4.602. PMID 10673877
- [Result] Adamik B, Kubler-Kielb J, Golebiowska B, Gamian A, Kubler A. Effect of sepsis and cardiac surgery with cardiopulmonary bypass on plasma level of nitric oxide metabolites, neopterin, and procalcitonin: correlation with mortality and postoperative complications. Intensive Care Med. 2000 Sep;26(9):1259-67. doi: 10.1007/s001340000610. PMID 11089751
- [Result] Fritz HG, Brandes H, Bredle DL, Bitterlich A, Vollandt R, Specht M, Franke UF, Wahlers T, Meier-Hellmann A. Post-operative hypoalbuminaemia and procalcitonin elevation for prediction of outcome in cardiopulmonary bypass surgery. Acta Anaesthesiol Scand. 2003 Nov;47(10):1276-83. doi: 10.1046/j.1399-6576.2003.00239.x. PMID 14616327
- [Result] Sablotzki A, Dehne MG, Friedrich I, Grond S, Zickmann B, Muhling J, Silber RE, Czeslick EG. Different expression of cytokines in survivors and non-survivors from MODS following cardiovascular surgery. Eur J Med Res. 2003 Feb 21;8(2):71-6. PMID 12626284
- [Result] Meisner M, Rauschmayer C, Schmidt J, Feyrer R, Cesnjevar R, Bredle D, Tschaikowsky K. Early increase of procalcitonin after cardiovascular surgery in patients with postoperative complications. Intensive Care Med. 2002 Aug;28(8):1094-102. doi: 10.1007/s00134-002-1392-5. Epub 2002 Jul 6. PMID 12185431
- [Result] Klingele M, Bomberg H, Schuster S, Schafers HJ, Groesdonk HV. Prognostic value of procalcitonin in patients after elective cardiac surgery: a prospective cohort study. Ann Intensive Care. 2016 Dec;6(1):116. doi: 10.1186/s13613-016-0215-8. Epub 2016 Nov 23. PMID 27878573